CLINICAL TRIAL: NCT00424944
Title: A Single Centre, Randomised Controlled Trial to Evaluate the Safety and Immunogenicity of Recombinant Lactococcus Lactis Hybrid GMZ 2 [GLURP + MSP 3] Blood Stage Malaria Vaccine Versus Rabies Vaccine in Healthy Gabonese Adult Volunteers
Brief Title: Safety of Recombinant Hybrid GMZ 2 [GLURP + MSP 3] Blood Stage Malaria Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Malaria Network Trust (Network)
Responsible Party: Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GMZ2_2_07
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Malaria
Keywords: Malaria; Vaccine; GMZ2; Safety; African; immunogenicity
MeSH Terms: conditions — Malaria | interventions — Malaria Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I, GMZ2 vaccine arm (Experimental): 20 volunteers will receive GMZ2 vaccine on days 0, 28, and 56
  Interventions: Biological: GMZ2 (malaria vaccine); Biological: GMZ2 malaria vaccine; Biological: Verorab vaccine
- II, Rabies vaccine arm (Active Comparator): 20 volunteers will receive standard vaccine against rabies on the similar schedule on days 0, 28, and 56
  Interventions: Biological: GMZ2 (malaria vaccine); Biological: Verorab vaccine

INTERVENTIONS:
Biological: GMZ2 (malaria vaccine) — 100 micrograms of GMZ2 in each vaccination
Biological: GMZ2 malaria vaccine — 100 micrograms of GMZ2
  Arms: I, GMZ2 vaccine arm
Biological: Verorab vaccine — Anti-rabies vaccine

SUMMARY:
The study aims to show that the candidate malaria vaccine GMZ2 is as safe as the already publicly used vaccine against rabies. 40 adult male Gabonese volunteers will be enrolled and randomly allocated to receive either malaria vaccine or rabies vaccine without the investigator or the participants knowing what they received. They will receive 3 doses each at one month intervals, and will be followed up for one year to evaluate safety parameters.

This is the first time this product will be tested in Africa

DETAILED DESCRIPTION:
Background. GMZ2 is a recombinant hybrid of the Glutamate Rich Protein (GLURP) and the Merozoite Surface Protein 3 (MSP 3).This product has been developed at Sate Serum Institute in Denmark and Bacth released by Henogen of Belgium. The phase Ia trial in malaria naive volunteers is currently ongoing in Germany, at Tuebingen University. This phase Ia trial will establish safety of the vaccine and also select the best dosage (10, 30 or 100 µg). The dosage with the best safety and immunogenicity profile will be recommended for the phase Ib trial in Gabon.

2. Study Design This will be a single center, randomized, blinded and controlled study involving 40 adult male volunteers. The entire study duration will be 16 months with each participant remaining 13 months in the study.There will be 15 scheduled hospital visits and 11 scheduled field worker home visits. The Rabies vaccine will be used as control vaccine.

3. Objectives:

- The primary objective of this trial to evaluate the safety of 3 doses of GMZ2 when administered on Days 0, 28 & 56, adjuvanted with aluminum hydroxide in healthy Gabonese adults.

- Secondary objectives include the following: (i). To assess the humoral response to the vaccine antigens GLURP and MSP3 by measuring the antibody response by ELISA and IFA.

(ii). To assess the cellular immune response by profiling the Th1/Th2-type cytokines after 24 and 48 hours stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male Gabonese 18-45 years inclusive at the time of screening
* Residing in Lambarene for the duration of the study
* Separate written informed consent obtained before screening and study start respectively
* Available to participate in follow-up for the duration of study (13 months)
* General good health based on history and clinical examination

Exclusion Criteria:

* Previous vaccination with a investigational vaccine or a rabies vaccine
* Use of a investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization, or planned use up to 30 days after the third immunization
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first immunization. This includes any dose level of oral steroids or inhaled steroids, but not topical steroids
* Confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Confirmed or suspected autoimmune disease
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine component
* History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care,or history of allergy to vaccines components
* History of splenectomy
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count 3.5-11/µL, absolute lymphocyte count 560-5280/µL, platelet count 120,000-400,000/µL, or hemoglobin 10.0-16.5g/dL).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period.
* Simultaneous participation in any other interventional clinical trial
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, malnutrition, or any other clinical findings that in the opinion of the clinical investigator may increase the risk of participating in the study
* Other condition that in the opinion of the clinical investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-07 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Local and systemic reactogenicity | 28 days following each immunization
Unsolicited adverse events | 1 year
Occurrence of serious adverse events | 1 year
Biological safety | 1 year

SECONDARY OUTCOMES:
Humoral immune response to GLURP and MSP 3 | 1 year
Cellural immune response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kremsner, MD, PhD, Study Director — Medical research Unit, Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon